CLINICAL TRIAL: NCT05281913
Title: A Web-based Psychoeducational Simulation Game for Remarried Adults - Study Protocol for a Randomized Controlled Trial.
Brief Title: Psychoeducational Simulation Game for Adults in Stepfamilies
Acronym: GSteps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FPCEUP/RH4
Record Dates: First submitted 2022-02-24; First posted 2022-03-16 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2022-11

CONDITIONS: Internet-Based Intervention; Remarriage
Keywords: remarriage; stepfamily; step-parenting; psychoeducation; web-based interventions; clinic interventions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A web-based Simulation Game concerning marital positive skills in remarriage, positive co-parenting strategies and positive stepparent-stepchild relationship skills.
  Interventions: Other: Psychoeducational Game
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Psychoeducational Game — Psychoeducational Game
  Arms: Intervention Group

SUMMARY:
Recent evidence has shown that intervention programs for remarried people are scarce.

Furthermore, from what is known, no specific intervention models (traditional or web-based) has yet been developed for remarried Portuguese population. This study evaluates the efficacy of a web-based Psychoeducational Simulation Game on marital adjustment on marital social skills, on remarriage beliefs, on parenting attitudes, and on the stepfamily functioning.

DETAILED DESCRIPTION:
This study will compare the efficacy of a Simulation Game Intervention versus control (no game) in remarried people that have (step)children. The participants will be randomized to the two groups. The Simulation Game contains three different modules to play: Module 1 - Conjugality (emotional divorce, financial issues, positive communication skills, conflict and stress management strategies, social support); Module 2 - Step-parenting (positive stepparent-stepchild relationships, development of relationships within stepfamily, step-parenting roles negotiation, stepfamily' unrealistic beliefs and develop share meaning); Module 3 - Co-parenting (positive co-parenting strategies and loyalty binds).

ELIGIBILITY:
Inclusion Criteria:

* Live in a Stepfamily
* Relationship length minimum of six months

Exclusion Criteria:

* Not having (step)children
* Not cohabiting with the spouse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Change in marital adjustment | T0 - before the intervention; T1 - immediately after intervention; T2 - one month later
  This measure is a self-rating questionnaire to assesses the quality of the dyadic relationship with three subscales: Consensus, Satisfaction and Cohesion.
Change in marital social skills | T0 - before the intervention; T1 - immediately after intervention; T2 - one month later
  This measure is a 32-item self-report measure that evaluates the frequency with which people present certain social skills in the context of their marital relationship.

SECONDARY OUTCOMES:
Change in Step-parenting Attitudes and Beliefs | T0 - before the intervention; T1 - immediately after intervention; T2 - one month later
  Seventeen items were used to rate the participants' step-parenting attitudes and beliefs addressed in the program content.
Change in Co-parenting Attitudes and Beliefs | T0 - before the intervention; T1 - immediately after intervention; T2 - one month later
  Nine items were used to rate the participants' co-parenting attitudes and beliefs addressed in the program content.
Change in remarriage Beliefs | T0 - before the intervention; T1 - immediately after intervention; T2 - one month later
  This measure is a self-rating questionnaire to assesses participants' unrealistic beliefs regarding remarriage and stepfamilies in general.
Change in stepfamily functioning | T0 - before the intervention; T1 - immediately after intervention; T2 - one month later
  This measure is a self-report questionnaire to provide an evaluation of family functioning with 5 items and three dimensions: Family strengths, Family communication and Family difficulties.

OTHER OUTCOMES:
Change in participants knowledge | T1 - immediately after intervention; T2 - one month later
  Twelve questions were specially elaborated for this study to assess the participants knowledge learned after the intervention.
Participants' Satisfaction with Intervention | T1 - immediately after intervention
  Self-report questionnaire to provide an evaluation of satisfaction with intervention through two dimensions: Usability and Content.

CONTACTS AND LOCATIONS:
Overall Officials: Carina Santos, MSc, Principal Investigator — Universidade do Porto
Locations (1):
- University of Porto, Faculty of Psychology and Educational and Education Sciences, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided